CLINICAL TRIAL: NCT03664999
Title: Dynamics of Serum Immunologic Markers Levels in During the Delivery and Possible Benefit for Obstetric Emergency Diagnostics
Brief Title: Serum Immunologic Markers Levels in During the Delivery
Acronym: DIMDOED
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FN Brno 2018/9
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Immunologic Markers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parturients physiologic pregnancy: Parturients undergoing caesarean delivery with physiologic pregnancy
  Interventions: Diagnostic Test: Blood sampling
- Parturients with risk pregnancy: Parturients undergoing caesarean with risk of complications (pre-eclampsia, HELLP syndrom, placenta praevia, placental abruption, IUGR, previous post partum hypotony).
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — differences between dynamics of the complement components C1 inhibitor, C1 inhibitor activity, C3, C4 during the labour in a group of women with physiologic pregnancy and in a group with a risk of complications (pre-eclampsia, HELLP syndrome, placenta praevia, placental abruption, IUGR, previous post partum hypotony).
  Other Names: Blood sample

SUMMARY:
This study aim to describe dynamics of immunologic markers C1 inhibitor, C3, C4 during the delivery in order to improve early diagnostics of obstetric emergencies, especially with immune etiology.

DETAILED DESCRIPTION:
Our prospective observational study will explore the differences between dynamics of the complement components C1 inhibitor, C1 inhibitor activity, C3, C4 during the labour in a group of women with physiologic pregnancy and in a group with a risk of complications (pre-eclampsia, HELLP syndrome, placenta praevia, placental abruption, IUGR, previous post partum hypotony).

We will focus on women undergoing the Caesarean delivery. We will also measure D vitamin levels and ACE levels and search for some contexts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing the Caesarean delivery
* Signed informed consent

Exclusion Criteria:

* Previous hepatitis or other hepatocyte damage

Ages: 15 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Parturients indicated for caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in levels of total C1 inhibitor | 30 minutes before and 30 minutes after delivery
  Chenge in levels of total C1 inhibitor
Change in levels of CRP levels | 30 minutes before and 30 minutes after delivery
  Change in levels of CRP levels
Change in levels of D vitamin levels | 30 minutes before and 30 minutes after delivery
  Change in levels of D vitamin levels and it's relationship to pre-eclampsia
Change in levels of ACE levels | 30 minutes before and 30 minutes after delivery
  Change in levels of ACE levels
Change of C1 inhibitor activity | 30 minutes before and 30 minutes after delivery
  Change of C1 inhibitor activity
Change in levels of total C3 | 30 minutes before and 30 minutes after delivery
  Change in levels of total C3
Change in levels of total C4 | 30 minutes before and 30 minutes after delivery
  Change in levels of total C4

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided